CLINICAL TRIAL: NCT02399319
Title: Prospective Randomized Comparison of Subcutaneous Internal Fixation ("INFIX") and Plating for Pelvic Ring Injuries With Symphysis Disruptions
Brief Title: Comparison of INFIX and Plating for Pelvic Ring Injuries With Symphysis Disruptions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principle Investigator left the institution
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1403899155
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2017-07

CONDITIONS: Anterior Pelvic Ring Injury With Symphysis Disruption
Keywords: anterior pelvic ring; symphysis disruption
MeSH Terms: interventions — Internal Fixators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Randomized to Internal Fixator (Experimental): Patient signed consent and agreed to have their treatment method randomized and the randomization system determined that their surgical intervention would be internal fixator.
  Interventions: Procedure: Internal Fixator
- Randomized to Symphyseal Plate (Experimental): Patient signed consent and agreed to have their treatment method randomized and the randomization system determined that their surgical intervention would be internal plating of the symphysis.
  Interventions: Procedure: Symphyseal Plate
- Observational - Internal Fixator (Active Comparator): Patient signed consent but did not want to randomize their procedure and the treating physician selected the internal fixator intervention based on their opinion of how best to treat the specific case.
  Interventions: Procedure: Internal Fixator
- Observational - Symphyseal Plate (Active Comparator): Patient signed consent but did not want to randomize their procedure and the treating physician selected internal plating of the symphysis based on their opinion of how best to treat the specific case.
  Interventions: Procedure: Symphyseal Plate

INTERVENTIONS:
Procedure: Internal Fixator — Internal fixator refers to pins usually inserted into the iliac bones and then connected together by clamps and bars that are inserted under the skin, internally.
  Arms: Observational - Internal Fixator; Randomized to Internal Fixator
Procedure: Symphyseal Plate — A plate that spans across the symphysis to maintain reduction and stability.
  Arms: Observational - Symphyseal Plate; Randomized to Symphyseal Plate

SUMMARY:
The purpose of this study is to compare subcutaneous internal fixation and open plating of the symphysis in patients with a disruption of the symphysis requiring stabilization.

DETAILED DESCRIPTION:
The aim of this study is to determine whether either one of the two procedures has significant advantages over the other. The null hypothesis of this study is that there is no difference between plating and subcutaneous internal fixation of symphysis disruptions with respect to primary and secondary outcomes. The study is a randomized trial with patients who sustained a symphysis disruption who will randomize to either closed reduction and subcutaneous internal fixation, or open reduction and plating of the symphysis. There will also be two observational arms of the study, patients who do not agree to randomization and will receive internal fixation according to the treating surgeon's discretion and patients with a symphysis disruption that do not require any form of anterior pelvic internal fixation based on the treating surgeon's opinion. Clinical assessments will occur at the time of hospital admission and at all post-operative follow-up intervals (2 weeks, 6 weeks, 3 months, 6months, 12 months, and 24 months).

ELIGIBILITY:
Inclusion Criteria:

* A symphysis disruption either in the coronal and/or sagittal plane on anterior-posterior , inlet and/or outlet pelvic radiographs
* Need for anterior pelvic ring stabilization
* Injury amenable to plating as well as subcutaneous internal fixation per the treating surgeon's opinion
* Patient was ambulatory prior to sustaining the injury
* Provision of informed consent by patient or proxy

Exclusion Criteria:

* Patients with a slim build with little subcutaneous fat who cannot be treated with a subcutaneous internal fixator based on the treating surgeon's opinion
* Patients who are deemed not likely to follow-up (e.g. patients who live more than 50 miles away and patients with no fixed address)
* Moderately or severely cognitively impaired patients
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07-21 (Actual); Study Completion 2016-07-21 (Actual)

PRIMARY OUTCOMES:
Functional Outcomes | 24 hours - 24 months
  The primary objective is to compare functional outcomes between subcutaneous internal fixation and symphyseal plating as measured by the PROMIS v1.2-Physical Function instrument.

SECONDARY OUTCOMES:
Compare the health-related quality of life and functional outcome scores | 24 hours - 24 months
  We will ask patients multiple questionnaires to assess their quality of life after surgery. These questionnaires include: PROMIS v1.1 - Pain Interference, PROMIS v1.2 - Mobility, PROMIS v1.0 - Global Satisfaction with Sex Life, PROMIS v1.0 - Depression, Majeed score, SF-12, VAS, patient satisfaction score, time to return to work, revision surgery, use of assistive walking devices, length of hospital stay, and for me, PROMIS v1.0 - Erectile Function.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zlowodzki, MD, Principal Investigator — Indiana University Health
Locations (1):
- Indiana University Health Methodist Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Dalal SA, Burgess AR, Siegel JH, Young JW, Brumback RJ, Poka A, Dunham CM, Gens D, Bathon H. Pelvic fracture in multiple trauma: classification by mechanism is key to pattern of organ injury, resuscitative requirements, and outcome. J Trauma. 1989 Jul;29(7):981-1000; discussion 1000-2. PMID 2746708
- [Background] Vallier HA, Cureton BA, Schubeck D, Wang XF. Functional outcomes in women after high-energy pelvic ring injury. J Orthop Trauma. 2012 May;26(5):296-301. doi: 10.1097/BOT.0b013e318221e94e. PMID 22337480
- [Background] Raman R, Roberts CS, Pape HC, Giannoudis PV. Implant retention and removal after internal fixation of the symphysis pubis. Injury. 2005 Jul;36(7):827-31. doi: 10.1016/j.injury.2004.11.012. Epub 2005 Feb 25. PMID 15949483
- [Background] Vallier HA, Cureton BA, Schubeck D. Pelvic ring injury is associated with sexual dysfunction in women. J Orthop Trauma. 2012 May;26(5):308-13. doi: 10.1097/BOT.0b013e31821d700e. PMID 22011632
- [Background] Vallier HA, Cureton BA, Schubeck D. Pregnancy outcomes after pelvic ring injury. J Orthop Trauma. 2012 May;26(5):302-7. doi: 10.1097/BOT.0b013e31822428c5. PMID 22048182
- [Background] Cole PA, Gauger EM, Anavian J, Ly TV, Morgan RA, Heddings AA. Anterior pelvic external fixator versus subcutaneous internal fixator in the treatment of anterior ring pelvic fractures. J Orthop Trauma. 2012 May;26(5):269-77. doi: 10.1097/BOT.0b013e3182410577. PMID 22357081
- [Background] Gardner MJ, Mehta S, Mirza A, Ricci WM. Anterior pelvic reduction and fixation using a subcutaneous internal fixator. J Orthop Trauma. 2012 May;26(5):314-21. doi: 10.1097/BOT.0b013e318220bb22. PMID 22048189
- [Background] Merriman DJ, Ricci WM, McAndrew CM, Gardner MJ. Is application of an internal anterior pelvic fixator anatomically feasible? Clin Orthop Relat Res. 2012 Aug;470(8):2111-5. doi: 10.1007/s11999-012-2287-6. PMID 22383020
- [Background] Moazzam C, Heddings AA, Moodie P, Cole PA. Anterior pelvic subcutaneous internal fixator application: an anatomic study. J Orthop Trauma. 2012 May;26(5):263-8. doi: 10.1097/BOT.0b013e31823e6b82. PMID 22337488
- [Background] Vaidya R, Kubiak EN, Bergin PF, Dombroski DG, Critchlow RJ, Sethi A, Starr AJ. Complications of anterior subcutaneous internal fixation for unstable pelvis fractures: a multicenter study. Clin Orthop Relat Res. 2012 Aug;470(8):2124-31. doi: 10.1007/s11999-011-2233-z. PMID 22219004
- [Background] Vaidya R, Colen R, Vigdorchik J, Tonnos F, Sethi A. Treatment of unstable pelvic ring injuries with an internal anterior fixator and posterior fixation: initial clinical series. J Orthop Trauma. 2012 Jan;26(1):1-8. doi: 10.1097/BOT.0b013e318233b8a7. PMID 22048183
- [Background] Majeed SA. External fixation of the injured pelvis. The functional outcome. J Bone Joint Surg Br. 1990 Jul;72(4):612-4. doi: 10.1302/0301-620X.72B4.2380212.
- [Background] Drummond M. Introducing economic and quality of life measurements into clinical studies. Ann Med. 2001 Jul;33(5):344-9. doi: 10.3109/07853890109002088. PMID 11491193
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] PELTIER LF. COMPLICATIONS ASSOCIATED WITH FRACTURES OF THE PELVIS. J Bone Joint Surg Am. 1965 Jul;47:1060-9. No abstract available. PMID 14318624
- [Background] Scaglione M, Parchi P, Digrandi G, Latessa M, Guido G. External fixation in pelvic fractures. Musculoskelet Surg. 2010 Nov;94(2):63-70. doi: 10.1007/s12306-010-0084-5. Epub 2010 Nov 18. PMID 21086087
- [Background] Pohlemann T, Bosch U, Gansslen A, Tscherne H. The Hannover experience in management of pelvic fractures. Clin Orthop Relat Res. 1994 Aug;(305):69-80. PMID 8050249
- [Background] Holstein JH, Pizanis A, Kohler D, Pohlemann T; Working Group Quality of Life After Pelvic Fractures. What are predictors for patients' quality of life after pelvic ring fractures? Clin Orthop Relat Res. 2013 Sep;471(9):2841-5. doi: 10.1007/s11999-013-2840-y. PMID 23408176
- [Background] Kabak S, Halici M, Tuncel M, Avsarogullari L, Baktir A, Basturk M. Functional outcome of open reduction and internal fixation for completely unstable pelvic ring fractures (type C): a report of 40 cases. J Orthop Trauma. 2003 Sep;17(8):555-62. doi: 10.1097/00005131-200309000-00003. PMID 14504576
- [Background] McCarthy ML, MacKenzie EJ, Bosse MJ, Copeland CE, Hash CS, Burgess AR. Functional status following orthopedic trauma in young women. J Trauma. 1995 Nov;39(5):828-36; discussion 836-7. doi: 10.1097/00005373-199511000-00005. PMID 7473997
- [Background] Mullis BH, Sagi HC. Minimum 1-year follow-up for patients with vertical shear sacroiliac joint dislocations treated with iliosacral screws: does joint ankylosis or anatomic reduction contribute to functional outcome? J Orthop Trauma. 2008 May-Jun;22(5):293-8. doi: 10.1097/BOT.0b013e31816b6b4e. PMID 18448980
- [Background] Oliver CW, Twaddle B, Agel J, Routt ML Jr. Outcome after pelvic ring fractures: evaluation using the medical outcomes short form SF-36. Injury. 1996 Nov;27(9):635-41. doi: 10.1016/s0020-1383(96)00100-3. PMID 9039360
- [Background] Suzuki T, Shindo M, Soma K, Minehara H, Nakamura K, Uchino M, Itoman M. Long-term functional outcome after unstable pelvic ring fracture. J Trauma. 2007 Oct;63(4):884-8. doi: 10.1097/01.ta.0000235888.90489.fc. PMID 18090021
- [Background] Matta JM. Indications for anterior fixation of pelvic fractures. Clin Orthop Relat Res. 1996 Aug;(329):88-96. doi: 10.1097/00003086-199608000-00011. PMID 8769439
- [Background] Matta JM, Saucedo T. Internal fixation of pelvic ring fractures. Clin Orthop Relat Res. 1989 May;(242):83-97. PMID 2706863
- [Background] Pohlemann T, Gansslen A, Schellwald O, Culemann U, Tscherne H. Outcome after pelvic ring injuries. Injury. 1996;27 Suppl 2:B31-8. PMID 8915200
- [Background] Tornetta P 3rd, Dickson K, Matta JM. Outcome of rotationally unstable pelvic ring injuries treated operatively. Clin Orthop Relat Res. 1996 Aug;(329):147-51. doi: 10.1097/00003086-199608000-00018. PMID 8769446
- [Background] Tornetta P 3rd, Matta JM. Outcome of operatively treated unstable posterior pelvic ring disruptions. Clin Orthop Relat Res. 1996 Aug;(329):186-93. doi: 10.1097/00003086-199608000-00022. PMID 8769450
- [Background] Lefaivre KA, Slobogean GP, Valeriote J, O'Brien PJ, Macadam SA. Reporting and interpretation of the functional outcomes after the surgical treatment of disruptions of the pelvic ring: a systematic review. J Bone Joint Surg Br. 2012 Apr;94(4):549-55. doi: 10.1302/0301-620X.94B4.27960. PMID 22434474
- [Background] Majeed SA. Grading the outcome of pelvic fractures. J Bone Joint Surg Br. 1989 Mar;71(2):304-6. doi: 10.1302/0301-620X.71B2.2925751.
- [Background] Lefaivre KA, Slobogean GP, Ngai JT, Broekhuyse HM, O'Brien PJ. What outcomes are important for patients after pelvic trauma? Subjective responses and psychometric analysis of three published pelvic-specific outcome instruments. J Orthop Trauma. 2014 Jan;28(1):23-7. doi: 10.1097/BOT.0b013e3182945fe9. PMID 23571293
- [Background] Sprague S, Leece P, Bhandari M, Tornetta P 3rd, Schemitsch E, Swiontkowski MF; S.P.R.I.N.T. Investigators. Limiting loss to follow-up in a multicenter randomized trial in orthopedic surgery. Control Clin Trials. 2003 Dec;24(6):719-25. doi: 10.1016/j.cct.2003.08.012. PMID 14662277
- See also: PROMIS outcome questionnaires — http://www.nihpromis.org/software/assessmentcenter